CLINICAL TRIAL: NCT04565054
Title: Adj. Dynamic Marker - Adjusted Personalized Therapy Comparing Abemaciclib Combined With Standard Adjuvant Endocrine Therapy Versus Standard Adjuvant Endocrine Therapy in (Clinical or Genomic) High Risk, HR+/HER2- EBC
Brief Title: Adjuvant Therapy With Abemaciclib + SOC ET vs. SOC ET in Clinical or Genomic High Risk, HR+/HER2- EBC
Acronym: ADAPTlate
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West German Study Group (Other)
Collaborators: Eli Lilly and Company (Industry); Genomic Health®, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSG-AM11 (ADAPTlate); 2019-001488-60 (EudraCT Number)
Record Dates: First submitted 2020-07-07; First posted 2020-09-25 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer Female
Keywords: early breast cancer; ADAPT; endocrine therapy; abemaciclib; high risk; HER2 negative; HR positive
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: multicenter, interventional, prospective, two-arm, randomized, open-label, controlled adjuvant, phase-III trial evaluating the efficacy and safety of abemaciclib with endocrine therapy (ET) versus standard-of-care endocrine therapy in early breast cancer (EBC) patients with molecular HR+/HER2- subtype.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Abemaciclib plus ET (Experimental): Abemaciclib 150 mg, 2 x daily, resulting in 300 mg/day, oral, 24 months plus endocrine treatment of physician´s choice
  Interventions: Drug: Abemaciclib 50 MG; 150mg 1-0-1 per os
- Standard-of-care ET (No Intervention): Standard-of-care ET according to clinical guidelines.
  Pre-/perimenopausal patients:
  * Either aromatase inhibitor + GnRH agonist
  * or Tamoxifen +/- GnRH-agonist (as per investigator´s decision) or
  Postmenopausal patients:
  * Either Aromatase inhibitor
  * or Tamoxifen OR

INTERVENTIONS:
Drug: Abemaciclib 50 MG; 150mg 1-0-1 per os — Experimental: Abemaciclib plus ET Abemaciclib 150 mg, 2 x daily, resulting in 300 mg/day, oral, 24 months plus endocrine treatment of physician´s choice
  Other Names: Verzenios
  Arms: Abemaciclib plus ET

SUMMARY:
Patients with breast cancer, who have completed first line therapy (e.g., radiotherapy, chemotherapy, surgery), and who have to be identified with having a high risk of recurrence of cancer, will be eligible for the study. This patient group is currently offered a standard of care chemotherapy plus endocrine therapy (ET). The study investigates whether the patient group with high-risk early breast cancer benefits from treatment with the medication abemaciclib in combination with ET compared to ET alone.

DETAILED DESCRIPTION:
The WSG ADAPT trial program is one of the first new generation trials addressing the issue of individualization of (neo)-adjuvant decision-making in early breast cancer (EBC) in a subtype-specific manner. The first WSG ADAPT umbrella trial (NCT01779206) aimed to establish early predictive molecular surrogate markers for response after a short 3-week induction treatment.

The goals of the WSG ADAPT trial program - early response assessment and subtype-specific therapy tailoring to those patients who are most likely to benefit - have contributed to the positive national and international feedback regarding the ADAPT-concept as a whole.

The aim of this ADAPTlate phase-III-trial is to gain further knowledge of the group of patients at intermediate to high risk for disease recurrence, who have completed definite locoregional therapy (with or without neoadjuvant or adjuvant chemotherapy). With ADAPTlate it is planned to investigate if the intermediate to high-risk patient group identified during the screening phase derives additional benefit from treatment with abemaciclib in combination with ET compared to ET alone.

ELIGIBILITY:
Inclusion Criteria:

A. Prior to REGISTRATION

1. Written informed consent prior to any study procedures (outcomes of standard-of-care procedures performed before signing of informed consent by the patient but within allowed screening period can be used for screening of patient). 2. Female. 3. ≥ 18 years of age. 4a. EITHER: (Post)menopausal status at the time of initiation of adjuvant study medication

* patient underwent bilateral oophorectomy, or
* age ≥ 60, or
* age < 60 and amenorrhea for 12 or more months (in the absence of chemotherapy, tamoxifen, or ovarian suppression) and/or FSH and estradiol in the postmenopausal range per local normal range.

  4b. OR: Pre-/perimenopausal patients:
* confirmed negative serum or urine pregnancy test (β-hCG) before starting study treatment, or
* patient has had a hysterectomy. 5. Histologically confirmed diagnosis(by local laboratory ) of estrogen-receptor positive and/or progesterone-receptor positive (>1% ) primary early breast cancer or local relapse. In case the receptor status from local pathology is unclear a central pathology review is obligatory. Results must be known prior to randomization.

  6. Patient has HER2-negative breast cancer defined as
* a negative in-situ hybridization test or an IHC status of 0, 1+, or 2+,
* if IHC is 2+, a negative in-situ hybridization (FISH, CISH, or SISH) test is required (based on the analyzed tissue sample at initial diagnosis by a local laboratory).

  7. Patients are eligible
* with completed (i.e., 5 years according to SoC), planned or ongoing adjuvant endocrine therapy, without any signs of distant relapse or secondary malignancy AND
* if primary diagnosis was 6 years or less before enrollment 8a. Intermediate to high clinical or genomic risk, defined as either one of the following criteria:
* c or p or ypN 2-3 with/without (neo)adjuvant chemotherapy;
* in patients with c/ypN0-1:
* non-pCR in patients with G3 or c/ypN1
* high biological risk defined as G3 with Ki-67 ≥40%
* or high genomic risk (RS>25 (known or Oncotype Dx® in screening phase) or another test)
* high CTS5 score or UICC stage IIb (clinical if neoadjuvant chemotherapy or pathological)

OR, if patients do not fulfill above criteria:

* patients ≤50 years old or pre-/perimenopausal and c or (y)pN1 disease (in particular if ET-non-response or no chemotherapy)
* patients >50 years old and postmenopausal and c or (y)pN1 with intermediate genomic risk (RS≥18) or non-low risk by another test

ET non-response definition:

Ki-67 post-treatment > 10% (central or local pathology value) OR 8b. Patients after isolated locoregional relapse with high-risk patterns (e.g., rpT2-3 or rpN1-3 or G3 or Ki-67 pre-treatment ≥20%), once surgery with free margins was completed Note: Inclusion is only possible for the first locoregional relapse removed by surgery (free margins) OR 8c. Patients with any high clinical risk at Investigator´s assessment but not fulfilling above criteria: consultation with sponsor required

B. Prior to RANDOMIZATION in the study 9. Completed primary therapy of breast cancer according to current guidelines, i.e., after (neo)adjuvant treatment, definite surgery and radiotherapy, if applicable.

10. No clinical evidence of distant metastasis (confirmation recommended prior to randomization by either combination of or either one of the following examinations: CT thorax / abdomen, chest X-ray, liver ultrasound, bone scan, PET-CT). 11. Patient has available tumor tissue from primary diagnostic biopsy. 12. No contraindication for adjuvant ET. 13. Eastern Cooperative Oncology Group (ECOG) performance status 0-1. 14. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

* absolute neutrophil count ≥ 1.5 × 109/L,
* platelets ≥ 100 × 109/L,
* hemoglobin ≥ 8.0 g/dL,
* total bilirubin ≤ 1.5 ULN, except for patients with Gilbert's Syndrome who may only be included if the total bilirubin is ≤ 2.0 × ULN or direct bilirubin within normal ranges,
* aspartate transaminase (AST) ≤ 3 × ULN,
* alanine transaminase (ALT) ≤ 3 × ULN,
* serum creatinine ≤ 1.5 x ULN. 15. Ability to swallow abemaciclib tablets or to administer other study medication, respectively.

  16. Ability to communicate with the investigator and comply with study procedures.

  17. Willing to receive therapy by clinical site, as required by the protocol.

Exclusion Criteria:

Patients eligible for inclusion in this study must not meet any of the following criteria:

1. Patient with distant metastases of breast cancer beyond regional lymph nodes.
2. Previously received CDK 4/6 inhibitor.
3. Patient with a known hypersensitivity to any of the excipients of abemaciclib or standard-of-care endocrine therapy.
4. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects.
5. Patient has not recovered from clinical and laboratory acute toxicities related to prior anticancer therapies to NCI CTCAE version 5.0 Grade ≤ 1 (polyneuropathy ≤ 2 is allowed).
6. Patient has a concurrent malignancy or non-breast malignancy within 5 years prior to randomization.
7. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small-bowel resection).
8. Patient has any active systemic bacterial infection (requiring intravenous antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment.
9. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator´s judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study, or compromise compliance with the protocol (e.g., interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea, etc.).
10. Patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest.
11. Patient is currently receiving any of the following substances, which cannot be discontinued 7 days prior to day 1 of study treatment:

    o concomitant medications and herbal supplements, that are strong inducers or inhibitors of CYP3A4.
12. Participation in a prior investigational study within 30 days prior to enrollment.
13. Not able to understand and to comply with study instructions and requirements.
14. Pregnant or nursing (lactating) woman.
15. Woman of child-bearing potential defined as woman physiologically capable of becoming pregnant, unless she is using highly effective methods of contraception during the study treatment and for 21 days after stopping the treatment:

    1. total abstinence (when this is in line with the preferred and usual lifestyle of the patient).
    2. female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy), total hysterectomy, or tubal ligation at least 6 weeks before taking study treatment.
    3. male partner sterilization (at least 6 months prior to study screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient.
    4. placement of an intrauterine device (IUD).
    5. use of condom + spermicide.
16. Use of oral (estrogen and progesterone), transdermal, injected, or implanted hormonal methods of contraception as well as hormonal replacement therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1260 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
invasive disease-free survival (iDFS) | at end of study, 3-6 years after start of study treatment
  superiority in invasive disease-free survival (iDFS) of abemaciclib + endocrine therapy vs. standard-of-care endocrine therapy in patients with HR+/HER2- high risk breast cancer.

SECONDARY OUTCOMES:
overall survival (OS) | at end of study, 3-6 years after start of treatment
  assessment of overall survival (OS) and distant DFS (dDFS) in both arms
differences in overall survival (OS) and dDFS | at end of study, 3-6 years after start of study treatment
  differences in overall survival (OS) and dDFS between arms
subgroup and multivariable survival analyses | at end of study, 3-6 years after start of study treatment
  subgroup and multivariable survival analyses
CNS metastases | at end of study, 3-6 years after start of study treatment
  occurrence of CNS metastases
EORTC QLQ-C30 | at end of study, on average 3-6 years after start of treatment
  quality of life (QoL)
EORTC QLQ-BR23 | at end of study, on average 3-6 years after start of treatment
  quality of life (QoL)
EQ-5D-5L | at end of study, on average 3-6 years after start of treatment
  quality of life (QoL)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Gluz, PD Dr. med., Principal Investigator — Westdeutsche Studiengruppe GmbH
Locations (85):
- Germany (70):
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau, Baden-Wurttemberg
  - SLK Kliniken Heilbronn Klinik für Gynäkologie und Geburtshilfe, Heilbronn, Baden-Wurttemberg
  - MVZ für Hämatologie und Onkologie, Ravensburg, Baden-Wurttemberg
  - Universitätsklinikum Ulm Frauenheilkunde, Geburtshilfe, Ulm, Baden-Wurttemberg
  - GRN-Klinik Weinheim Gynäkologie und Geburtshilfe, Weinheim, Baden-Wurttemberg
  - Klinikum Mittelbaden Balg, Baden-Baden, Baden-Würtemberg
  - Universitätsklinikum Tübingen Department für Frauengesundheit, Brustzentrum, Tübingen, Baden-Wüttenburg
  - Haematologie-Onkologie im Zentrum MVZ GmbH, Augsburg, Bavaria
  - Klinikum der Universität München Campus Großhadern Frauenheilunde und Geburtsklinik, Munich, Bavaria
  - Medizinisches Zentrum für Hämatologie und Onkologie München MVZ GmbH, Munich, Bavaria
  - Rotkreuzkliniken München, Interdisziplinbäres Brustzentrum, München, Bavaria
  - Hämatologisch-Onkologische Schwerpunktpraxis Würzburg & Kitzingen, Würzburg, Bavaria
  - Medizinische Universität Lausitz - Carl-Thiem Frauenklinik, Cottbus, Brandenburg
  - Klinikum Ernst von Bergmann gGmbH Brustzentrum, Potsdam, Brandenburg
  - Centrum für Hämatologie und Onkologie, Frankfurt a.M., Hesse
  - Brustzentrum, Elisabeth-Krankenhaus gGmbH, Kassel, Hesse
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Langen, Hesse
  - St. Josefs-Hospital Wiesbaden GmbH Ambulanz der Frauenklinik, Brustzentrum, Wiesbaden, Hesse
  - Studien GbR Braunschweig Dr. Lorenz/Dr. Kreiss-Sender, Braunschweig, Lower Saxony
  - MVZ II der Niels Stensen Kliniken Onkologie u. Hämatologie, Georgsmarienhütte, Lower Saxony
  - MVZ Onkologische Kooperation Harz (GbR), Goslar, Lower Saxony
  - Diakovere Krankenhaus gGmbH Henriettenstift Frauenklinik, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover Frauenheilkunde, Hanover, Lower Saxony
  - MVM Medizinische Verwaltungs und Managementgesellschaft mbH, Leer, Lower Saxony
  - Pius-Hospital Oldenburg Hämatologie, Onkologie, Oldenburg, Lower Saxony
  - Klinikum Südstadt Rostock Frauenklinik, Rostock, Mecklenburg-Vorpommern
  - Stiftung Katholisches BrustCentrum Marienhospital, Aachen, North Rhine-Westphalia
  - Uniklinik RWTH Aachen Gynäkologie und Geburtsmedizin, Aachen, North Rhine-Westphalia
  - Evangelisches Krankenhaus Bergisch Gladbach gGmbH Brustzentrum,, Bergisch Gladbach, North Rhine-Westphalia
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld, North Rhine-Westphalia
  - Gynäkologisches Zentrum Bonn PD Dr. med. Christian Kurbacher, Bonn, North Rhine-Westphalia
  - GYNONOVA GbR Schwerpunktpraxis für gynäkologische Onkologie, Cologne, North Rhine-Westphalia
  - St. Elisabeth-Krankenhaus GmbH, Brustzentrum - Senologie, Cologne, North Rhine-Westphalia
  - Kliniken der Stadt Köln Krankenhaus Köln-Holweide Medizinische Klinik Brustzentrum, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf Frauenheilkunde und Geburtshilfe, Düsseldorf, North Rhine-Westphalia
  - MVZ Medical Center Duesseldorf GmbH Luisenkrankenhaus Brustzentrum, Düsseldorf, North Rhine-Westphalia
  - St.-Antonius-Hospital Eschweiler Hämatologie/Onkologie, Eschweiler, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Klinik für Senologie/Interdisziplinäres Brustzentrum, Essen, North Rhine-Westphalia
  - Universitätsklinikum Essen Frauenheilkunde und Geburtshilfe, Essen, North Rhine-Westphalia
  - Onkodok GmbH Onkologische Schwerpunktpraxis, Gütersloh, North Rhine-Westphalia
  - Praxisgemeinschaft Gynäkologische Onkologie & Spezielle Operative Gynäkologie, Hildesheim, North Rhine-Westphalia
  - Zentrum für ambulante gynäkologisch Onkologie (ZAGO), Krefeld, North Rhine-Westphalia
  - Städtisches Klinikum Lüneburg Frauenklinik, Lüneburg, North Rhine-Westphalia
  - Johannes Wesling Klinikum Minden Innere Medizin, Hämatologie, Onkologie, Minden, North Rhine-Westphalia
  - Brustzentrum Niederrhein, im ev. Krankenhaus Bethesda, Mönchengladbach, North Rhine-Westphalia
  - Universitätsklinikum Münster AöR Brustzentrum, Münster, North Rhine-Westphalia
  - Marien Krankenhaus Schwerte MKS St. Paulus GmbH, Schwerte, North Rhine-Westphalia
  - Praxisnetz Hämatologie / internistische Onkologie, Troisdorf, North Rhine-Westphalia
  - Christliches Klinikum Unna Mitte Gynäkologie und Geburtshilfe, Unna, North Rhine-Westphalia
  - Marien Hospital Witten Brustzentrum, Witten, North Rhine-Westphalia
  - Helios Universitätsklinikum Wuppertal Landesfrauenklinik, Wuppertal, North Rhine-Westphalia
  - Praxisklinik für Hämatologie und Onkologie Koblenz, Koblenz, Rhineland-Palatinate
  - Klinikum Mutterhaus der Borromäerinnen Innere Medizin 1, Trier, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes Klinik für Frauenheilkunde, Homburg (Saar), Saarland
  - Caritas Traegergesellschaft Saarbruecken mbH (CTS) Frauenklinik, Saarbrücken, Saarland
  - Klinikum Chemnitz Frauenheilkunde und Geburtshilfe, Chemnitz, Saxony
  - Onkozentrum Dresden/Freiberg/Meißen, Dresden, Saxony
  - Gemeinschaftspraxis Dr. med. Johannes Mohm, Dr. med. Virág Siklaky, Stefanie Mann Onkopraxis Dresden, Dresden, Saxony
  - Universitätsklinikum Leipzig, Klinik und Poliklinik für Frauenheilkunde, Leipzig, Saxony
  - Klinikum St. Georg Gynäkologie und Geburtshilfe, Leipzig, Saxony
  - Klinikum Obergöltzsch Brustzentrum Vogtland, Rodewisch, Saxony
  - Universitätsklinikum Halle (UKH), Universitätsklinik und Poliklinik für Gynäkologie, Halle, Saxony-Anhalt
  - Klinikum Magdeburg Frauenheilkunde und Geburtshilfe, Magdeburg, Saxony-Anhalt
  - Johanniter Krankenhaus Frauenklinik, Stendal, Saxony-Anhalt
  - MediOnko-Institut GbR Praxiskliik Krebsheilkunde für Frauen/Brustzentrum, Berlin
  - Praxis für gynäkologische Onkologie im Brustzentrum City am Sankt Gertrauden KH, Berlin
  - HELIOS Klinikum Berlin-Buch GmbH, Berlin
  - Onkologisch-Hämatologische Schwerpunktpraxis, Bremen
  - AGAPLESION Diakonie-Klinikum Hamburg Gyn. Studienambulanz, Hamburg
  - Mammazentrum Hamburg MVZ GbR, Hamburg
- Poland (3):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Uniwersytet Jagiellonski Collegium Medicum Szpital Uniwersytecki w Krakowie - Klinika Onkologii, Krakow
  - MSCM Cancer Center and Institute of Oncology Department of Breast Cancer and Reconstructive Surgery, Warsaw
- Spain (12):
  - Hospital Universitari Son Espases, Palma, Mallorca
  - Hospital Vall Hebron - Vall Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital Universitario San Pedro De Alcantara, Cáceres
  - Hospital Universitario de Vinalopo, Elche
  - Hospital Beata Maria Ana, Madrid
  - Althaia Xarxa Assistencia, Manresa
  - Hospital Regional Universitario Malaga, Málaga
  - Hospital Universitario De Navarra, Pamplona
  - Hospital Universitario San Juan De Alicante, Sant Joan d'Alacant
  - Complejo Hospitalario Universitario Santiago de Compostela, Santiago de Compostela
  - Hospital Quironsalud Sagrado Corazon, Seville
  - Consorcio Hospital General Universitario De Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No